CLINICAL TRIAL: NCT07300956
Title: Comparing Medication Treatments for Neurodevelopmental Differences in Young Children on Rates of Beneficial Response
Brief Title: Treating Young Children With Attention Deficit Hyperactivity Disorder
Acronym: TYCA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Children's Hospital of Philadelphia (Other); Developmental Behavioral Pediatrics Research Network (Unknown); Boston Children's Hospital, Boston, MA, USA (Other); Children's Mercy Hospital Kansas City (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Tanya Froehlich, MD, Division Director, Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPS-2024C2-39495
Record Dates: First submitted 2025-12-22; First posted 2025-12-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: Attention-Deficit/Hyperactivity Disorder; Methylphenidate; Guanfacine; Preschool Children; Comparative Effectiveness; Prospective Study
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine; Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Guanfacine (Active Comparator): After engaging in behavioral therapy, participants randomized to this group will be prescribed Guanfacine. The child's prescribing clinician will determine the form and dose of Guanfacine that the child receives.
  Interventions: Drug: Guanfacine (GUA)
- Methylphenidate (Active Comparator): After engaging in behavioral therapy, participants randomized to this group will be prescribed Methylphenidate. The child's prescribing clinician will determine the form and dose of Methylphenidate that the child receives.
  Interventions: Drug: Methylphenidate (MPH)

INTERVENTIONS:
Drug: Guanfacine (GUA) — After engaging in behavioral therapy, participants randomized into this group participants will be prescribed Guanfacine. Each child's prescribing clinician determines the form and dose of guanfacine that the child receives.
  Guanfacine (GUA) medication brand names include: Intuniv, Tenex, guanfacine hydrochloride- extended release, guanfacine hydrochloride- immediate release
  Arms: Guanfacine
Drug: Methylphenidate (MPH) — Participants randomized into this group will be prescribed Methylphenidate. Each child's prescribing clinician determines the form and dose of methylphenidate that the child receives.
  Methylphenidate (MPH) medication brand names include: Adhansia XR, Aptensio XR, Azstarys, Concerta, Cotempla XR-ODT, Daytrana, Focalin, Focalin XR, Jornay PM. Metadate CD, Methylin (liquid), Relexxii, Ritalin, Ritalin LA, Quillichew ER, Quillivant XR (liquid), methylphenidate hydrochloride- extended release, methylphenidate hydrochloride- immediate release
  Arms: Methylphenidate

SUMMARY:
This project will evaluate the effectiveness of Methylphenidate versus Guanfacine in treating Attention-Deficit/Hyperactivity Disorder (ADHD) in children aged 3 through 5 years (inclusive), as measured by clinician rating of global improvement.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is one of the most common neurodevelopmental disorders, affecting 2-3% of U.S. children under 6 (also called preschool-age children. Preschool Attention-Deficit/Hyperactivity Disorder is linked to difficulties in school or daycare, with friendships and family relationships, and accidental injuries. Behavioral therapy is recommended as the first step in treating preschool-age Attention-Deficit/Hyperactivity Disorder. However, for some children, behavior therapy is not enough. For these children, medication may also be needed to treat their Attention-Deficit/Hyperactivity Disorder.

The most common medications used to treat Attention-Deficit/Hyperactivity Disorder in preschool-age children are Methylphenidate and Guanfacine. Currently, there is not enough research to help families and doctors choose between these two medications when treating this age group. This research study will fill this gap by directly comparing the benefits and side effects of Methylphenidate and Guanfacine for treating Attention-Deficit/Hyperactivity Disorder in this age group, giving families and clinicians the information they need to make evidence-based treatment choices.

The main goal of this study is to compare the effectiveness of Methylphenidate and Guanfacine in children ages 3-5, focusing on clinically meaningful improvement in overall functioning. Clinicians will measure the child's improvement using the Clinical Global Impressions scale.

There are also secondary goals in this study. One of those secondary goals is to understand how acceptable and tolerable each of these medications is, from the family perspective and the clinician perspective. This will be learned in a few ways. It will be measured through how long participants choose to stay on the medication and through surveys from caregivers about medication side effects (Pittsburgh Side Effect Rating Scale) at the beginning of the study and again 4, 8, 12, and 16 weeks after starting medication.

The other secondary goals are to understand if medication choice impacts a child and their family in other ways (e.g. behavioral symptoms, parenting stress) and learn about any factors that may influence a child's response to medication (e.g. age, initial symptoms). This information will primarily come from caregiver surveys (Parenting Stress Index, Vanderbilt Attention-Deficit/Hyperactivity Disorder Parent Rating Scales, Affective Reactivity Index). If the caregiver agrees, and the child has a teacher, their teacher will also complete surveys (Vanderbilt Attention-Deficit/Hyperactivity Disorder Teacher Rating Scales, Affective Reactivity Index). The Vanderbilt Attention-Deficit/Hyperactivity Disorder Rating Scales are completed at the beginning of the study and again 4, 8, 12, and 16 weeks after starting medication. The Parenting Stress Index and Affective Reactivity Index are completed at the beginning of the study and again 8 and 16 weeks after starting medication.

Caregivers and their child will be required to attend 3 in person visits (before starting medication and again 8 weeks and 16 weeks after starting medication. At these visits, a study doctor will measure the child's height, weight, blood pressure, and heart rate to make sure that the medication is safe to start or continue. The other 3 visits with study doctors can be in-person or online. If a teacher is completing study surveys, they will all be available through a secure, online platform.

This study uses a randomization to compare the effectiveness of Methylphenidate and Guanfacine in preschool-age children with Attention-Deficit/Hyperactivity Disorder, including how side effects may differ.

This study aims to provide evidence-based guidance on using Methylphenidate and Guanfacine in treating Attention-Deficit/Hyperactivity Disorder in preschool-age children. Evidence about each medicine's effectiveness in this age group will help families and clinicians make more informed decisions when treating preschool-age children with Attention-Deficit/Hyperactivity Disorder.

This research study is being co-designed with parents, clinicians, and health systems stakeholders. Working with these stakeholders helps ensure that the research will be practical for families, clinicians, and health systems. Caregivers of children with Attention-Deficit/Hyperactivity Disorder, who are 3-5 (inclusive) will be recruited to participate. Across the United States, 5 total sites will participate to enroll a total of 370 children in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 3 to 5 years of age, inclusive (e.g. children age 5 years, 11 months are eligible).
2. Child has a confirmed diagnosis of moderate or severe Attention-Deficit/Hyperactivity Disorder (diagnostic code: F90.9) based on Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5) criteria, review of supportive evidence (caregiver interview, behavioral observations, Vanderbilt Attention-Deficit/Hyperactivity Disorder Rating Scale results, any school or daycare information provided by caregiver).
3. Clinician-rated Clinical Global Impairment-Severity (see description below) rating of ≥4 (denoting moderate or greater impairment due to their Attention-Deficit/Hyperactivity Disorder symptoms).
4. The child's clinician and caretakers have decided on or are considering initiating drug therapy (with either Methylphenidate or Guanfacine).
5. Primary language is English or Spanish.

Exclusion Criteria:

1. History of taking Methylphenidate or Guanfacine. Prior use of other Attention-Deficit/Hyperactivity Disorder medications or other psychotropic medications is allowed.
2. Current use of other Attention-Deficit/Hyperactivity Disorder medications (e.g., amphetamines), other psychotropic medications (e.g., atypical antipsychotics or serotonin reuptake inhibitors), or centrally active depressants (such as phenothiazines, barbiturates, or benzodiazepines)
3. Electronic Health Record documentation of moderate to severe global developmental delay (F88) or intellectual disability (F70), or a score of <55 on the Vineland Adaptive Behavior Scales-3.
4. Medical contraindications to taking Methylphenidate or Guanfacine, including cardiac risk factors (e.g. known structural cardiac abnormalities, cardiomyopathy, serious cardiac arrhythmias, coronary artery disease, or other serious cardiac disease), increased intraocular pressure, glaucoma, verbal tics, Tourette's Syndrome, psychosis

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 370 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression-Improvement | From enrollment to the end of the 16-week medication treatment.
  The Clinical Global Impression-Improvement scale is a seven-point rating tool that evaluates how a participant's Attention-Deficit/Hyperactivity Disorder symptoms have changed since their baseline measurement. Although this scale can be used for other mental health conditions, in this study it is applied specifically to Attention-Deficit/Hyperactivity Disorder. A score of "1" indicates "very much improved," while a score of "7" indicates "very much worse." Higher scores reflect a worse outcome.

SECONDARY OUTCOMES:
Medication discontinuation within 16 weeks | From medication randomization assignment to the end of the 16-week medication treatment.
  The percent of participants who discontinue medication prior to 16 weeks will be measured to assess treatment acceptability.
Vanderbilt Attention-Deficit/Hyperactivity Disorder Parent Rating Scales | From enrollment to the end of the 16-week medication treatment.
  This caregiver-completed questionnaire includes 55 items across three sections. The first section contains 18 Attention-Deficit/Hyperactivity Disorder symptom items rated on a three-point scale from "Never" (0) to "Very Often" (3), with Attention-Deficit/Hyperactivity Disorder total symptom scores ranging from a minimum of 0 to a maximum of 54. The second section contains 29 items related to behavioral and mental health comorbidity symptoms (e.g., oppositional defiant, disordered conduct, anxiety, and mood symptoms) rated on a three-point scale from "Never" (0) to "Very Often" (3), with comorbidity total symptom scores ranging from a minimum of 0 to a maximum of 87. The third section includes eight performance/impairment-related items rated on a five-point scale from "Excellent" (1) to "Problematic" (5), with performance/impairment total scores ranging from 8 to 40. On all sections, higher scores indicate more severe symptoms and/or greater impairment.
Vanderbilt Attention-Deficit/Hyperactivity Disorder Teacher Rating Scales | From enrollment to the end of the 16-week medication treatment.
  This measure, completed by teachers (if applicable), includes 43 items divided into three sections. The first section contains 18 Attention-Deficit/Hyperactivity Disorder symptoms items rated on a three-point scale from "Never" (0) to "Very Often" (3), with Attention-Deficit/Hyperactivity Disorder total symptom scores ranging from a minimum of 0 to a maximum of 54. The second section contains 17 items related to behavioral and mental health comorbidity symptoms (e.g., oppositional defiant, disordered conduct, anxiety, and mood symptoms) rated on a three-point scale from "Never" (0) to "Very Often" (3), with comorbidity total symptom scores ranging from 0 51. The third section includes eight performance/impairment-related items rated on a five-point scale from "Excellent" (1) to "Problematic" (5), with performance/impairment total scores ranging from 8 to 40. On all sections, higher scores indicate more severe symptoms and/or greater impairment.
Parenting Stress Index Short Form | From enrollment to the end of the 16-week medication treatment.
  Caregivers will complete the Parenting Stress Index Short Form, which consists of 36 items. Each item is rated on a five-point scale ranging from 1= "Strongly Disagree" to 5= "Strongly Agree." Total scores can range from 36 to 180, with higher scores indicating greater levels of parenting stress.
Affective Reactivity Index - Caregiver | From enrollment to the end of the 16-week medication treatment.
  This measure, completed by caregivers, includes 7 items. For each item, the caregiver responds by answering 0="Not True," 1="Somewhat True," or 2="Certainly True." Total scores range from 0 to 14. Higher scores indicate higher levels of irritability, whereas lower scores indicate lower levels of irritability.
Affective Reactivity Index - Teacher | From enrollment to the end of the 16-week medication treatment.
  This measure, completed by teachers (if applicable), includes 7 items. For each item, teachers respond by answering 0="Not True," 1="Somewhat True," or 2="Certainly True." Total scores range from 0 to 14. Higher scores indicate higher levels of irritability, whereas lower scores indicate lower levels of irritability.
Pittsburgh Side Effects Rating Scale | From enrollment to the end of the 16-week medication treatment.
  The Pittsburgh Side Effects Rating Scale will be completed by caregivers and will measure safety and tolerability. This version of the scale has been adapted to include one additional item related to daytime sleepiness, a known side effect of Guanfacine, resulting in a total of 14 items. Each item is rated on a scale from 0 to 3, where 0 means the side effect is not present, 1 means the side effect is mild, 2 means the side effect is moderate, and 3 means the side effect is severe. Total scores range from 0 to 42, with 0 indicating no side effect symptoms and higher scores indicating more/worse side effects.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford Medicine Children's Health, Palo Alto, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
At this time, we do not plan to share individual participant data from this study. Our Institutional Review Board approval is contingent upon maintaining participant privacy and confidentiality, and sharing individual-level data would not be consistent with these requirements. While we may share aggregated, de-identified summary findings in publications or presentations, we cannot share any data that could potentially be linked back to individual participants. Only summary-level results will be made publicly available through publications and ClinicalTrials.gov.